CLINICAL TRIAL: NCT02519920
Title: Lower Fluorescein Sodium Dose on Confocal Laser Endoscopy Image Quality and Yellow Discoloration of the Skin
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Vice president of Qilu Hospital, Shandong University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 2015SDU-QILU-G08
Record Dates: First submitted 2015-08-03; First posted 2015-08-11 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-09

CONDITIONS: Image Quality; Skin Discoloration
MeSH Terms: interventions — Fluorescein

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- group 1 (Experimental): This group patients were given dosages of fluorescein sodium 0.01ml/kg intravenous administration.
  Interventions: Drug: fluorescein sodium 0.01ml/kg
- group 2 (Experimental): This group patients were given dosages of fluorescein sodium 0.02ml/kg intravenous administration.
  Interventions: Drug: fluorescein sodium 0.02ml/kg
- group 3 (Experimental): This group patients were given dosages of fluorescein sodium 0.05ml/kg intravenous administration.
  Interventions: Drug: fluorescein sodium 0.05ml/kg
- group 4 (Active Comparator): This group patients were given dosages of fluorescein sodium 0.1ml/kg intravenous administration.
  Interventions: Drug: fluorescein sodium 0.1ml/kg

INTERVENTIONS:
Drug: fluorescein sodium 0.01ml/kg — fluorescein Sodium Dose of 0.01ml/kg on confocal laser endoscopy image quality and yellow discoloration of the skin
  Arms: group 1
Drug: fluorescein sodium 0.02ml/kg — fluorescein Sodium Dose of 0.02ml/kg on confocal laser endoscopy image quality and yellow discoloration of the skin
  Arms: group 2
Drug: fluorescein sodium 0.05ml/kg — fluorescein Sodium Dose of 0.05ml/kg on confocal laser endoscopy image quality and yellow discoloration of the skin
  Arms: group 3
Drug: fluorescein sodium 0.1ml/kg — fluorescein Sodium Dose of 0.1ml/kg on confocal laser endoscopy image quality and yellow discoloration of the skin
  Arms: group 4

SUMMARY:
This study was to test an appropriate dose of fluorescein sodium which can provide high image quality to ensure endoscopy examination and have no yellow dye in the skin by a randomized blinded controlled trial.

DETAILED DESCRIPTION:
Fluorescein sodium is one of the commonly used staining agents in confocal laser endoscopy, a device for in vivo real-time histological observation of the gastrointestinal mucosa. The conventional intravenous dosage of fluorescein sodium is in the range of 5ml to 10ml of 10% fluorescein. Image quality can be guaranteed with this range of fluorescein sodium, but yellow discoloration of the skin seriously influences daily life. This study was to test whether a lower dose of fluorescein sodium, which has minimal discoloration of skin, can provide satisfied image quality by a randomized blinded controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Only those with normal mucosa and minor gastritis from 18 were included.
* patients with aged 18 years to 80 years
* patients with normal mucosa and minor gastritis
* willing to provide informed consent

Exclusion Criteria:

* serious coagulopathy dysfunction, severe cardiopulmonary disease, bronchial asthma, liver and kidney dysfunction, allergy to fluorescein, pregnancy women or breast feeding.
* patients with peptic ulcer, gastric cancer, remnant stomach, acute serious gastritis were also excluded.
* unwilling to provide informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2015-04; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Different ratios of high resolution CLE images among four different fluorescein sodium dose groups(0.01ml/kg,0.02ml/kg,0.05ml/kg,0.1ml/kg) | six months

SECONDARY OUTCOMES:
Different degrees of skin yellow dye of patients in four different fluorescein sodium dose groups(0.01ml/kg,0.02ml/kg,0.05ml/kg,0.1ml/kg) | six months

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, PhD.MD, Study Director — Department of Gastroenterology,Qilu Hospital,Shandong University
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China